CLINICAL TRIAL: NCT02264119
Title: Influence of 40 mg Pantoprazole Per Day on the Pharmacokinetics of Fradafiban After Multiple Oral Doses of 20 mg Lefradafiban Tid as Acid Free Tablet and Sachet Over 5 Days in Healthy Subjects. A 4-way Crossover Randomized Open Trial.
Brief Title: Influence of Pantoprazole on the Pharmacokinetics of Fradafiban After Multiple Oral Doses of Lefradafiban in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 509.119
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — lefradafiban; Pantoprazole

ARMS (4):
- Lefradafiban tablet with Pantoprazole (Experimental)
  Interventions: Drug: Lefradafiban tablet; Drug: Pantoprazole tablet
- Lefradafiban tablet without Pantoprazole (Active Comparator)
  Interventions: Drug: Lefradafiban tablet
- Lefradafiban double chamber sachet with Pantoprazole (Experimental)
  Interventions: Drug: Pantoprazole tablet; Device: Lefradafiban double chamber sachet
- Lefradafiban double chamber sachet without Pantoprazole (Active Comparator)
  Interventions: Device: Lefradafiban double chamber sachet

INTERVENTIONS:
Drug: Lefradafiban tablet
  Arms: Lefradafiban tablet with Pantoprazole; Lefradafiban tablet without Pantoprazole
Drug: Pantoprazole tablet
  Arms: Lefradafiban double chamber sachet with Pantoprazole; Lefradafiban tablet with Pantoprazole
Device: Lefradafiban double chamber sachet
  Arms: Lefradafiban double chamber sachet with Pantoprazole; Lefradafiban double chamber sachet without Pantoprazole

SUMMARY:
Study to assess the absorption of 20 mg Lefradafiban in two formulations, each under physiological conditions and with 40 mg Pantoprazole

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 60 years, planned stratification: age < 40 years (4 subjects) and ≥ 40 years (8 subjects)
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Drug abuse
* Alcohol abuse (> 60 g/day)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Excessive physical activities within 5 days prior to administration or during the trial
* Blood donation within 1 month prior to administration or during the trial
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders
* Chronic or relevant acute infections
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* History of

  * Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * Any bleeding disorder including prolonged or habitual bleeding
  * Other hematologic disease
  * Cerebral bleeding (e.g. after a car accident)
* Recent surgical procedures
* Thrombocytes < 150000/µ
* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Any laboratory value outside the clinically accepted reference range
* Other disease or abnormality of clinical relevance

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1998-04; Primary Completion 1998-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state, 13th dosing interval (AUCss,13) | Up to 168 hours after first drug administration
Maximum concentration of the analyte in plasma at steady state, 13th dosing interval (Cmax,ss,13) | Up to 168 hours after first drug administration
Pre-dose concentration of the analyte in plasma at steady state, 13th dosing interval (Cpre,ss,13) | Up to 168 hours after first drug administration
Amount of the analyte eliminated unchanged in the urine per dosing interval (Ae% (i=1,...,13)) | Up to 168 hours after first drug administration

SECONDARY OUTCOMES:
Pre-dose concentration lf the analyte in plasma for the i-th dosing interval (Cpre,i (i=1,4,7,10,11,12)) | Up to 168 hours after first drug administration
Plasma concentration of the analyte at 2 hours post-dose for the i-th dosing interval (C2h,i (i=10,11,12)) | up to 2 hours after each dosing interval
Terminal half life of the analyte in plasma (t1/2) | Up to 168 hours after first drug administration
Percent swing of peak/trough concentrations of the analyte in plasma for the i-th dosing interval (%Swing,i) | Up to 168 hours after first drug administration
  Calculated: (C2h,i - Cpre,i) / Cpre,i * 100% (i=10,11,12)
Percent peak-trough fluctuation for the 13th dosing interval (%PTF13) | Up to 168 hours after first drug administration
  Calculated: (Cmax,ss,13 - Cpre,ss,13) * 8h / AUCss,13 * 100%)
Percent fluctuation of area under the plasma concentration-time curve (AUCfluc,13) | Up to 168 hours after first drug administration
  Calculated: (AUCabove,13 - AUCbelow,13) / AUCabove,13
Fibrinogen receptor occupancy levels | Up to 168 hours after first drug administration
Number of subjects with adverse events | Up to 3 days after last drug administration
Number of subjects with clinically significant findings in vital signs | Up to 3 days after last drug administration
  systolic and diastolic blood pressure, pulse rate
Number of subjects with clinically significant findings in laboratory tests | Up to 3 days after last drug administration